CLINICAL TRIAL: NCT00561639
Title: Benefit of Septifast Multiplex PCR in the Etiologic Diagnosis and Therapeutic Approach for Onco-hematology Patients Presenting Sepsis
Acronym: SEPTIFAST
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: TIMSIT, University Hospital, Grenoble
Other Study IDs: 2007-A01053-50
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Hematologic Diseases; Sepsis
Keywords: sepsis; immunosuppressed; multiplex PCR; diagnosis; therapeutic
MeSH Terms: conditions — Hematologic Diseases; Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum tube will routinely be kept in the serum bank for subsequent analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A SpetiFast multiplex PCR kit has recently been placed on the market witch can evidence the DNA of 90% of micro-organisms (bacteria and fungus) implicated in sepsis. However, the clinical impact of being able to detect the DNA of these various agents is unknown. We propose to assess the benefit to patient care of the SeptiFast multiples PCR by answering three questions : 1/in patients with septic immunosuppression, does this kit evidence etiologic agents not revealed by classical methods? 2/Does the use of PCR results permit different diagnostic hypotheses to be considered? 3/Does having the SeptiFast results entail changes to the therapeutic plan?

DETAILED DESCRIPTION:
This study has double purpose :

1. To compare the results obtained from the SeptiFast system with the results from classical microbiological sampling, in particular hemoculture, for immunosuppressed patients presenting sepsis.
2. To perform a blind assessment of the benefit of septiFast care of these patients.

ELIGIBILITY:
Inclusion Criteria:

All patients with onco-hematologic or cancerous pathology, or hematologic disease with chemotherapy and/or radiotherapy and/or some other immunosuppressant treatment in progress presenting an infection requiring hospitalisation and meeting the following criteria:

* Sepsis (at least one of the following signs):

  * Fever > 38.2°C or hypothermia < 36°C
  * FO120 min
  * PA<120 mmHg (or 50 mmHg reduction in base numbers)
  * Respiratory F > 30/min
  * Confusion
  * Hyperleucocytosis (>12 G/l) or leucopenia (<4 G/l)
  * C-Reactive protein > 40
* With or without organ dysfunction as defined by :

  * Hypoxia (PaO2/FiO2<300mmHg)
  * Oliguria (urine deficiency<0.5 ml/kg/h in probed patient)
  * Creatinine > 200umol/l
  * INR>1.5 or TCA>2 X control in the absence of anticoagulant treatment
  * Platelets < 100 G/l
  * Bilirubin > 35 umol/l
  * Lactatemia > 2 mmol/l
  * Arterial hypotension (PAS<90mmHg, or PAM<70mmHg or reduction of more than 40 mmHG if known hypertension)

Exclusion Criteria:

* Minor patient
* Pregnancy
* A patient cannot be included again within 15 days of his/her preceding inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with onco-hematologic or cancerous pathology, or hematologic disease with chemotherapy and/or radiotherapy and/or some other immunosuppressant treatment in progress presenting an infection requiring hospitalisation and meeting the following criteria : Sepsis and with or without organ dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2007-12; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT Jean-François, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France